CLINICAL TRIAL: NCT01999036
Title: Save Hearts in Arizona Registry and Education (SHARE) Project
Acronym: SHARE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Arizona (Other)
Collaborators: Arizona Department of Health Services (Other Government)
Responsible Party: Principal Investigator, Bentley J. Bobrow, Professor of Emergency Medicine, University of Arizona
Other Study IDs: 11-0046
Record Dates: First submitted 2013-10-18; First posted 2013-12-03 (Estimated); Last update posted 2018-05-09 (Actual); Status verified 2018-05

CONDITIONS: Out-of-hospital Cardiac Arrest
Keywords: cardiac arrest, CPR, resuscitation
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest; Heart Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Resuscitation of OHCA: Resuscitation of out-of-hospital cardiac arrest

SUMMARY:
Evaluation of the impact of bystander CPR, prehospital resuscitation protocols, and hospital post-resuscitation protocols for out-of-hospital cardiac arrest patients in the state of Arizona.

ELIGIBILITY:
Inclusion Criteria:

* Out of Hospital Cardiac Arrest (loss of spontaneous circulation and EMS attempted resuscitation)

Exclusion Criteria:

* Do Not Resuscitate

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Out-of-hospital cardiac arrest patients on which resuscitation was attempted by Emergency Medical Services in the state of Arizona
Sampling Method: Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2004-11; Primary Completion 2020-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Survival to hospital discharge | Upon hospital discharge and annually up to 5 years
  Patients will be followed for the duration of hospital stay. The average time from admission to either discharge or death is expected to be approximately 2 weeks.

SECONDARY OUTCOMES:
Emergency Medical Services Cardiopulmonary Resuscitation (CPR) quality | Prehospital resuscitation
  Chest compression depth, rate, recoil, fraction. Patients will be followed for the duration of prehospital resuscitation. The average timeframe is expected to be approximately 15 minutes.

OTHER OUTCOMES:
Frequency and Quality of Telephone Cardiopulmonary Resuscitation (CPR) | During 9-1-1 call
  The average 9-1-1 call is expected to be approximately 8 minutes.
Proportion of out-of-hospital cardiac arrest patients receiving bystander Cardiopulmonary Resuscitation (CPR) | Time of cardiac arrest to EMS arrival
  Type of bystander Cardiopulmonary Resuscitation (CPR) given, if any. The average length of time between cardiac arrest and EMS arrival is expected to be approximately 10 minutes.
Proportion of out-of-hospital cardiac arrest patients transported to a recognized Cardiac Receiving Center | Emergency Medical Services (EMS) patient encounter
  The average patient encounter timeframe is expected to be approximately 15 minutes.
Proportion of out-of-hospital cardiac arrest patients receiving Guideline post-arrest care | Hospital admission to hospital discharge/death
  The average time from hospital admission to either discharge or death is expected to be approximately 2 weeks.
Post cardiac arrest care process | Hospital admission to hospital discharge/death
  Post arrest care measures include therapeutic hypothermia and percutaneous coronary intervention. Patients will be followed for the duration of their hospital stay. The average time from hospital admission to either discharge or death is expected to be approximately 2 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Multiple Locations, Arizona, United States

REFERENCES:
- [Derived] Irisawa T, Vadeboncoeur TF, Karamooz M, Mullins M, Chikani V, Spaite DW, Bobrow BJ. Duration of Coma in Out-of-Hospital Cardiac Arrest Survivors Treated With Targeted Temperature Management. Ann Emerg Med. 2017 Jan;69(1):36-43. doi: 10.1016/j.annemergmed.2016.04.021. Epub 2016 May 27. PMID 27238827